CLINICAL TRIAL: NCT00713115
Title: Prospective Randonmized Comparison of Needlescopic Versus Conventional Laparoscopic Adrenalectomy for Benign Adrenal Tumors Less Than 5 cm in Diameter
Brief Title: Prospective Randonmized Comparison of Needlescopic Versus Conventional Laparoscopic Adrenalectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shih-Chieh Chueh, Department of Urology, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200803040R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-06

CONDITIONS: Adrenal Tumors
Keywords: laparoscopy, needlescopy, adrenalectomy
MeSH Terms: conditions — Adrenal Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: needlescopic adrenalectomy and laparoscopic adrenalectomy — Needlescopic instruments, defined as those with a diameter of no more than 3 mm. They result in smaller incisions than conventional 5- to 12-mm instruments.
  Other Names: Miniscopic

SUMMARY:
The study is a prospective radonmized comparison between needlescopic adrenalectomy and conventional laparoscopic adrenalectomy for benign adrenal tumors less than 5 cm. The operative success rate, operative time, intraoperative blood loss, intraoperative or postoperative complication, postoperative pain, postoperative hospital stay, convalescence, and wound cosmesis were compared.

DETAILED DESCRIPTION:
Needlescopic instruments, defined as those with a diameter of no more than 3 mm. They result in smaller incisions than conventional 5- to 12-mm instruments, and thus better cosmesis. It may further reduce postoperative pain, hospital stay, and recovery time.

All operations were performed with the lateral transperitoneal approach. A 12-mm port was created near the umbilicus for a 30-degree telescope, and another two(for left lesions) or three (for right lesions) 2-mm working ports (Tyco Healthcare, Norwalk, Connecticut, USA) were created along the ipsilateral subcostal region. Careful dissection was done with the use of a 2-mm hook or scissors electrocoagulator. The adrenal vein of the lesion side was isolated and controlled with a 2-mm mini-bipolar coagulation apparatus (Tyco Healthcare) for a long segment. The vein was then transected closer to the adrenal gland, leaving the coagulated stump at the renal vein or vena cava as long as possible, even when a short right adrenal vein was encountered. Then the adrenal gland with the tumor was dissected from its surrounding tissues after several tiny vessels were transected with the needlescopic instruments mentioned above. The specimen was put into a retrieval bag and removed through the umbilical port.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Benign Adrenal Tumors

Exclusion Criteria:

* Suspected adrenal malignancy clinically
* Bilateral adrenal disease
* Pregnant female

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Operative time, blood loss, intraoperative and postoperative complication, pain score, convalescence, cosmesis | 1 month

SECONDARY OUTCOMES:
cost | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Chieh Chueh, MD. PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Liao CH, Lai MK, Li HY, Chen SC, Chueh SC. Laparoscopic adrenalectomy using needlescopic instruments for adrenal tumors less than 5cm in 112 cases. Eur Urol. 2008 Sep;54(3):640-6. doi: 10.1016/j.eururo.2007.12.028. Epub 2007 Dec 26. PMID 18164803